CLINICAL TRIAL: NCT01953263
Title: A Phase 1 Study of Human Muscle Fiber Fragment (MFF) Treatment for Urinary Incontinence
Brief Title: Muscle Fiber Fragment Treatment for Urinary Incontinence
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Wake Forest University (Other)
Responsible Party: Sponsor
Organization: Wake Forest University Health Sciences (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRB00025341
Record Dates: First submitted 2013-09-25; First posted 2013-09-30 (Estimated); Last update posted 2026-01-28 (Actual); Status verified 2025-05

CONDITIONS: Urinary Incontinence
Keywords: urinary incontinence, muscle fibers
MeSH Terms: conditions — Urinary Incontinence

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Autologous Muscle Fiber Fragments (Experimental): Autologous Muscle Fiber Fragments administered via a single,direct injection into the bladder neck sphincter region
  Interventions: Other: Autologous Muscle Fiber Fragments

INTERVENTIONS:
Other: Autologous Muscle Fiber Fragments — Autologous muscle fiber fragments administered via a single direct injection into the bladder neck sphincter region

SUMMARY:
This study is designed to evaluate the safety of autologous muscle fiber fragments for the treatment of urinary incontinence due to incompetent outlet (bladder neck/urethra).

DETAILED DESCRIPTION:
Eligible subjects with a diagnosis of urinary incontinence who give consent to take part will undergo a biopsy of the muscle from the inner thigh under anesthesia. During the same procedure, muscle fiber fragments will be obtained from the sample and then immediately delivered via target injected into the bladder neck sphincter region using an endoscopic needle via cystoscope or under ultrasound guidance. All subjects will be followed at 1 week, 6 weeks, 3 months, 6 months and 12 months post-treatment injection.

ELIGIBILITY:
Inclusion Criteria:

* Adult female patients who are not pregnant or lactating/breast-feeding and must be either not sexually active, surgically sterilized, or must be practicing an effective method of birth control as determined by the investigator
* Patients between the ages of 18 and 75 years
* Patients with positive diagnosis of urinary incontinence due to sphincter insufficiency caused by acquired (e.g., stress urinary incontinence) and/or congenital conditions.
* Patients with cystometric capacity of bladder > 100 ml
* Patients with normal renal function
* Patients with a history of primary incontinence

Exclusion Criteria:

* Patients with a history of hypercontractile bladder, non-compliant bladder, hydronephrosis or neurogenic bladder
* Patients with an active urinary tract infection as evidenced by positive urine culture
* Patients who are taking medication that affect urination such as prescription drugs, over-the-counter drugs, or dietary supplements, including herbal supplements and those taken with teas
* Patients requiring concomitant use of or treatment with immunosuppressive agents
* Patients with a history of systemic conditions, including but not limited to HIV, diabetes and chronic liver disease (including Hepatitis B or C), that the Investigator believes may jeopardize the safety of the patient to participate in the study
* Patients with evidence or diagnosis of any primary muscle disease or coagulation disorder (including concomitant anti-coagulation therapy)
* Patients who have been treated with any other investigational drug or participated in any investigational study within 30 days prior to enrollment in this study
* Patients who have been treated with any cellular therapy within 12 months prior to enrollment in this study
* Patients with urinary incontinence other than the categories being investigated
* Patients with significant (>grade 2) pelvic organ prolapse
* Patients with vaginal prolapse beyond introitus
* Patients with neurological disorders
* Patients with abnormal bladder capacity (i.e., less than 100 cc)
* Patients with abnormal urologic conditions, including post-void residual, urethral stricture and bladder neck contracture, spastic bladder, vesicoureteral reflux, bladder stones, bladder tumors, hydronephrosis, other renal impairment

Ages: 18 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2016-01; Primary Completion 2027-12 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
Incidence of treatment-related serious adverse events | 12 months
  the subject/biopsy/treatment sites will be monitored for signs of bleeding, infections, continued pain, prolonged hospitalization

SECONDARY OUTCOMES:
Change in Incontinence Assessment by Pad Test | baseline, 3, 6, and 12 months post-treatment
  Subjects will undergo 1 hour and 24 hour Pad Tests (pads are weighed) at baseline, 3, 6 and 12 months post treatment

OTHER OUTCOMES:
Change in number of incontinence episodes and pads used per day | baseline, 3, 6 and 12 months post-treatment
  voiding diaries and pads used each day will be compared to baseline

CONTACTS AND LOCATIONS:
Overall Officials: Gopal Badlani, MD, Principal Investigator — Wake Forest School of Medicine, Dept. of Urology
Locations (1):
- Wake Forest Urology Clinic, Winston-Salem, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No